CLINICAL TRIAL: NCT04690361
Title: Monitoring the EMG Activity and Investigating the Relation Between Occlusal Contact Areas and Occlusal Loads During Light or Heavy Occlusal Forces
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202008002RINA
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Bite Force, EMG
Keywords: occlusal contact,occlusal force,Electromyography,Dental PreScale System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Inappropriate occlusal contact may affect the long-term prognosis of prosthodontic rehabilitation. It is suggested to design light or without occlusal contact on implant prostheses when the patient bites with light force, and normal occlusal contact when the patient bites with heavy force. The concept of this "implant-protective occlusion" is based on the difference of movement between implants and natural teeth. However, how much force generated during a light bite or a heavy bite is not clearly defined in the literature. Traditional methods to evaluate the occlusal contacts between antagonist teeth such as wax, silicone, occlusal paper, and occlusal foil cannot evaluate the occlusal force. Recently, modern digital occlusion analysis systems (T-Scan, Dental Prescale II) can evaluate occlusal force on almost normal intermaxillary relation. The objects of this investigation are: (1) to evaluate the effect of difference occlusal forces on the number, distribution and size of occlusal contacts examined by 8μm occlusal foil and Dental Prescale II System (DPS); (2) to analyze the relation between EMG activity and occlusal forces and to identify the magnitude of light and heavy bite force the patients may exert during occlusal examination; (3) to compare the results between habitual chewing side and the other side. Twenty-four subjects will be included in this study. With EMG biofeedback, the subjects will exert 35%、70%、100% of maximum contraction EMG of clenching and the subjects' occlusal contacts will be tested with the 8μm occlusal foil and DPS. Each condition will be tested three times. The subjects will chew gums to confirm their habitual chewing side after the occlusal tests. Numbers, distribution, and size of occlusal contacts will be analyzed and compared. This study may identify the magnitude of perceptual light and heavy occlusal forces and the maximum occlusal force. The results are helpful for setting up the protocol and strategy of occlusal adjustment and to prevent biomechanical complications of dental prostheses.

ELIGIBILITY:
Inclusive criteria:

* full dentition except third molar
* class I occlusion at bilateral canines and first molars (Angle's classification)
* healthy periodontal condition
* can sign consent

Exclusive criteria:

-history of temporomandibular disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. healthy subject of dental patient at NTUH
  2. dental students
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-19 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The relation between occlusal force and EMG data | immediately after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: TongMei Wang, PHD, Principal Investigator — School of Dentistry, National Taiwan University College of Medicine.
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan